CLINICAL TRIAL: NCT06672263
Title: Phase I Clinical Trial to Evaluate the Safety and Tolerability of TQB3911 Tablets in Patients With BCR::ABL Fusion Gene Positive Leukemia
Brief Title: A Clinical Trial to Evaluate the Safety and Tolerability of TQB3911 Tablets in Patients With BCR::ABL Fusion Gene Positive Leukemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3911-I-01
Record Dates: First submitted 2024-10-27; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-07

CONDITIONS: Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3911 tablets (Experimental): Once a day for 28 days as a treatment cycle
  Interventions: Drug: TQB3911 tablets

INTERVENTIONS:
Drug: TQB3911 tablets — TQB3911 is a small molecule BCR::ABL1 allosteric inhibitor. By occupying the myristyl binding site, TQB3911 recovers the inhibition of BCR::ABL1 fusion protein kinase activity, and ultimately inhibits the proliferation of tumor cells.

SUMMARY:
Phase I clinical trial to explore the safety, tolerability, and initial efficacy of TQB3911 tablets in BCR::ABL fusion gene positive leukemia.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed the informed consent, and had good compliance;
* Age: ≥18 years old (when signing the informed consent); Eastern Cooperative Oncology Group Performance Status (ECOG PS) score: 0-2; Expected survival of more than 3 months;
* During the screening period, the patients were identified as Chronic myelogenous leukemia-Chronic phase (CML-CP) or accelerated phase (AP) patients by bone marrow cell morphological examination, molecular biological examination or cytogenetic examination;
* Chronic myelogenous leukemia (CML) patients who are intolerant to Tyrosine kinase inhibitors (TKI) drugs or whose therapeutic effect is not satisfactory (that is, the therapeutic response evaluation result is failure)
* The main organs function well
* Female subjects of reproductive age should agree to use contraceptives (such as Iuds, contraceptives, or condoms) during the study period and for 6 months after the end of the study; Have a negative serum pregnancy test within 7 days prior to study enrollment and must be a non-lactating subject; Male subjects should agree to use avoidance during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

* Had or was currently suffering from other malignant tumors within 5 years before the first medication
* Combined with active central nervous system leukemia
* Major surgical treatment and significant traumatic injury were received within 28 days before the start of study treatment
* Previous history of myocardial infarction, pulmonary hypertension, or angina pectoris within 3 months before the first medication, or clinically significant arrhythmias such as ventricular tachycardia, complete left bundle branch block, and high atrioventricular block
* Acute pancreatitis and a history of chronic pancreatitis within 12 months before the first medication
* History of interstitial lung disease, radiation pneumonia requiring steroid treatment, or drug-related pneumonia
* Patients with CML-CP who have achieved complete cytogenetic response (CCyR)
* Received live attenuated vaccine within 4 weeks before the first dose, or planned to receive live attenuated vaccine during study participation
* Use of drugs that may have caused QT prolongation or tip torsical tachycardia in the 7 days prior to initial administration, or continuation of these medications during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase II recommended doses (RP2D) | Baseline up to 24 months
  The dosage of drug therapy recommended for use in the second phase of clinical trials (i.e., phase II clinical trials).
Dose-limiting toxicity (DLT) | Up to 1 month
  Adverse events that meet the protocol definition of dose-limiting toxic event timing were evaluated according to the Common Terminology Criteria for Adverse Events 5.0.

SECONDARY OUTCOMES:
Incidence and severity of adverse event (AE) and serious adverse event (SAE), and abnormal laboratory test indicators | From the signing of informed consent for administration to 28 days after the last administration/start of the new antitumor therapy (whichever occurs first).
  Incidence and severity of AE and SAE, and abnormal laboratory test indicators
Peak time | Single dose on days 1 to 3, day 8 of cycle 1, day 15 of cycle 1, day 22 of cycle 1, and day 2 to day 1, each cycle is 28 days.
  Time to peak blood concentration after a single dose
C-QT Research | Single dose: 1 hour, 0.5 hour, 10 minutes before dose and 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 12 hours, 24 hours after dose.
  Effect of TQB3911 on QTcF interval in subjects
Platelet count | For the first six weeks, the assessment was weekly. Starting at week 6, assessments were performed at week 8 and every 4 weeks (±7 days) thereafter
  Hematologic remission of subjects during treatment
The proportion of Philadelphia chromosomes in the metaphase of bone marrow cells | They were evaluated every 12 weeks (±7 days) for 96 weeks and every 24 weeks (±7 days) after 96 weeks
  Cytogenetic remission of subjects during treatment
Molecular reaction | They were evaluated every 12 weeks (±7 days) for 96 weeks and every 24 weeks (±7 days) after 96 weeks
  Molecular remission of subjects during treatment
Progression free survival | They were evaluated every 12 weeks (±7 days) for 96 weeks and every 24 weeks (±7 days) after 96 weeks
  The period of time between the subject's treatment and the observation of disease progression or death from any cause
Overall survival | They were evaluated every 12 weeks (±7 days) for 96 weeks and every 24 weeks (±7 days) after 96 weeks
  The time from the subject's initiation of treatment or diagnosis until the patient's death from any cause
Peak concentration Cmax | Single dose on days 1 to 3, day 8 of cycle 1, day 15 of cycle 1, day 22 of cycle 1, and day 2 to day 1, each cycle is 28 days.
  After a single dose, the highest point of the drug-time curve is called the peak concentration
Plasma elimination half-life t1/2 | Single dose on days 1 to 3, day 8 of cycle 1, day 15 of cycle 1, day 22 of cycle 1, and day 2 to day 1, each cycle is 28 days.
  The amount of time it takes for the concentration of the drug in the blood, or the amount of drug in the body, to drop to about half of its original level.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang